CLINICAL TRIAL: NCT06602401
Title: Investigation of Functional Parameters: Relationships Between Bimanual Coordination, Proprioception, Manuel Dexterity, and Strength
Brief Title: Investigation of Functional Parameters
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Collaborators: Ali ZORLULAR (Unknown); Tuğçe ÇOBAN (Unknown); Ahmet GÖKKURT (Unknown); Zeynep EMİR (Unknown); Nevin ATALAY GÜZEL (Unknown); Deran OSKAY (Unknown)
Responsible Party: Principal Investigator, Barış SEVEN, Ph.D. research assistant, Gazi University
Other Study IDs: 4
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Grip; Pinch; Strength; Wrist; Dexterity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this cross-sectional study is to investigate the relationships between grip/pinch strengths, wrist flexion-extension strengths, wrist proprioception, manual dexterity, and bimanual coordination in healthy volunteers. The hypotheses are:

H0: There is no relationship between grip/pinch strengths, wrist flexion-extension strengths, wrist proprioception, manual dexterity, and bimanual coordination.

H1: There is a relationship between grip/pinch strengths, wrist flexion-extension strengths, wrist proprioception, manual dexterity, and bimanual coordination.

Within the scope of the study, the participants' active joint position sense (AJPS) and flexion-extension strengths of the wrist were assessed using an isokinetic dynamometer. Additionally, grip strength, key pinch, tip pinch, and palmar pinch strengths were evaluated using a dynamometer. The Purdue Pegboard Test was used to assess manual dexterity and bimanual coordination.

ELIGIBILITY:
Inclusion Criteria:

After providing detailed information about the research, individuals who agreed to participate were included in the study.

Exclusion Criteria:

Individuals who had undergone surgery or trauma in the upper extremity, had fractures or acute orthopedic injuries, had a history of neuromuscular diseases or congenital anomalies, had skin infections, or other conditions that could affect the assessment within the past 6 months were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: No specific age or disease/injury group is targeted. The study was conducted with healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
The Purdue Pegboard Test was used to assess bimanual coordination. | Participants will be evaluated only once.
  In the Purdue Pegboard test, participants, seated in front of the test board, were asked to placed pins into the holes on both sides of the board simultaneously with both hands as many pins as possible within 30 seconds. The total number of pins placed was recorded as the score for bimanual coordination.
The Purdue Pegboard Test was used to assess manual dexterity. | Participants will be evaluated only once.
  In the Purdue Pegboard test, participants, seated in front of the test board, were first asked to use their dominant hand to pick up pins from the dominant side and place them into the holes on the same side, from top to bottom. They were instructed to place as many pins as possible within 30 seconds. The number of pins placed was recorded as the score for dominant hand manual dexterity. The same test was then conducted for the nondominant side.
The active joint position sense was assessed using an isokinetic dynamometer. | Participants will be evaluated only once.
  For the assessment of wrist proprioception, an isokinetic dynamometer with demonstrated reliability [Cybex NORM®, Humac, CA, USA] was used.
  Wrist proprioception was assessed by Active Joint Position Sense (AJPS) measurement. During the test, participants wore eye masks. For the AJPS assessment, the target angle was set at 30° extension, which is the functional position of the wrist. Participants were asked to actively move their wrist from the neutral position to the 30° extension and hold this position for 5 seconds. This trial was repeated three times. Participants were then asked to find the target angle three times. The amount of error between the target angle and the achieved angle was used to define the accuracy of the active joint position sense. The arithmetic mean of these three measurements was calculated and recorded.
The flexion-extension strengths of the wrist were assessed using an isokinetic dynamometer. | Participants will be evaluated only once.
  Wrist flexion and extension strengths were also evaluated using the Cybex isokinetic dynamometer. These strength assessments were conducted in the same position and range of motion as the proprioception evaluations. Before starting the measurements, participants were informed about the test. At the beginning of the test, three practice trials were performed. The concentric-concentric strength measurement was conducted with an angular velocity of 60°/s for 5 repetitions. A 20-second rest period was allowed between the practice and test trials. The peak torque parameters for wrist flexion and extension in both wrists were measured.
  Assessments began with the dominant side. Subsequently, the same measurements were repeated on the other extremity by adjusting the position of the dynamometer and chair. The device was calibrated before the participants were evaluated. All measurements were conducted by the same person to prevent inter-rater variability.
Grip and pinch strengths were measured using a digital dynamometer. | Participants will be evaluated only once.
  The assessment of gross grip strength was performed using a digital dynamometer (J-Tech Commender Grip Track). Measurements were taken with the participant seated, the elbow flexed at 90 degrees, the wrist in up to 30 degrees of extension, and the forearm in a neutral rotation position. The dynamometer's grip width was set to the second level. Maximum grip force was measured by having the participant squeeze as hard as possible three times, and the arithmetic mean of these three measurements was calculated. Key pinch, palmar pinch, and tip pinch strength measurements were conducted using a pinch gauge (Baseline Mechanical Pinch Gauge, 60 lb) in the same position and with the same measurement technique as the gross grip strength assessment. All evaluation protocols were established according to the recommendations of the American Society of Hand Therapists.

CONTACTS AND LOCATIONS:
Locations (1):
- Barış SEVEN, Izmir, Çiğli, Turkey (Türkiye)